CLINICAL TRIAL: NCT00004686
Title: Phase II Randomized Study of Glucocorticoids With or Without Methotrexate for Treatment of Giant Cell Arteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13298; CCF-RPC-4586; CCF-FDR001040; DPT-32-0-48
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Giant Cell Arteritis
Keywords: cardiovascular and respiratory diseases; giant cell arteritis; rare disease
MeSH Terms: conditions — Giant Cell Arteritis; Respiratory Tract Diseases; Rare Diseases | interventions — Methotrexate; Prednisone

INTERVENTIONS:
Drug: methotrexate
Drug: prednisone

SUMMARY:
OBJECTIVES: I. Compare the long term outcomes in patients with giant cell arteritis after glucocorticoid treatment with or without methotrexate.

II. Compare remission relapse rates in these patients after glucocorticoid therapy with or without methotrexate.

III. Determine whether adjunctive use of methotrexate lowers cumulative dose and duration of glucocorticoid therapy and whether there is less treatment related morbidity and mortality.

IV. Demonstrate the feasibility of long term, double blind, placebo controlled, randomized, multicenter trials for treatment of systemic vasculitides.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, multicenter study. Patients are randomized into initial therapy with prednisone plus weekly placebo or prednisone plus weekly oral methotrexate. Patients who do not respond to treatment within 5 days are taken off study. If methotrexate toxicity dose not occur after 2 weeks, methotrexate is increased by one tablet per week until a maximum tolerated dose (MTD) is achieved. The MTD of methotrexate or the matching placebo dose is continued for 12 months in the absence of toxicity. Once 12 continuous months of remission are achieved, methotrexate or placebo is tapered to discontinuation.

Patients are followed for 1-6 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of giant cell arteritis (GCA) by at least one of the following:

* Temporal artery biopsy confirming GCA Symptoms of GCA (including new onset (within 6 months) symptoms of headaches, tenderness of the scalp or the temporal arteries, visual loss due to retinal ischemic optic neuropathy or otherwise unexplained tongue or jaw pain) and an aortic angiogram that revealed stenotic and/or aneurysmal disease of the aorta and its principal branches
* Symptoms of polymyalgia rheumatica plus ischemic optic neuropathy, newly identified tenderness over a temporal artery, or new onset of tongue or jaw pain

Westergren erythrocyte sedimentation rate of at least 40 nm in one hour

--Prior/Concurrent Therapy--

Endocrine therapy: No greater than 20 days since initiation of prednisone therapy

Other: No concurrent sulfa drugs or nonsteroidal antiinflammatory drugs

--Patient Characteristics--

Hematopoietic:

* WBC at least 4,000/mm3
* Platelet count at least 120,000/mm3
* No acute or chronic liver disease

Hepatic:

* Alkaline phosphatase no greater than 2 times upper limit of normal
* No other reproducible abnormal liver function test

Renal: Creatinine less than 2.0 mg/dL

Other:

* HIV negative
* No symptomatic peptic ulcer disease within the last 3 months
* Hepatitis B or C antigen negative
* No alcohol use in excess of 2 ounces of 100 proof liquor or 1 beer or its equivalent per week
* No insulin dependent diabetes mellitus plus morbid obesity (greater than 33% over ideal body weight)
* No recently (less than 6 months) diagnosed malignancy
* Not pregnant or nursing
* Adequate contraception required of all fertile patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1994-02; Study Completion 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Gary Stuart Hoffman, Study Chair — The Cleveland Clinic